CLINICAL TRIAL: NCT01449448
Title: A Double-blind Randomized Controlled Trial Comparing the Effects of Subacromial Injection With Corticosteroid Versus NSAID in Patients With Shoulder Impingement Syndrome
Brief Title: Subacromial Injection With Corticosteroid Versus Nonsteroidal Anti-inflammatory Drugs (NSAID) in Shoulder Impingement Syndrome
Acronym: NSAID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI didn't have time to finish approval process
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: impingement
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Subacromial Impingement Syndrome; Subacromial Bursitis
Keywords: pain relief; Hypermobility, Joint; increased strength; increased patient satisfaction
MeSH Terms: conditions — Shoulder Impingement Syndrome; Joint Instability | interventions — Ketorolac; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSAID (Experimental): Test Group: This group was given subacromial injections of Ketorolac.
  Interventions: Drug: Ketorolac
- Steroid (Active Comparator): This group was given a subacromial injection triamcinolone.
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Ketorolac — Subacromial injection
  Arms: NSAID
Drug: Triamcinolone — Subacromial Injection
  Arms: Steroid

SUMMARY:
Injection with corticosteroid is one of the most common non-operative interventions in the treatment of subacromial impingement; however, its use is limited by its potential side effects (e.g. tendon rupture, subcutaneous atrophy, articular cartilage changes). The objective of this study was to compare the efficacy of subacromial injection of triamcinolone compared to injection of ketorolac. Thirty-two patients diagnosed with external shoulder impingement syndrome were included in this double-blinded randomized controlled clinical trial. Each patient was randomized into the Steroid group or NSAID group.

DETAILED DESCRIPTION:
After a single injection into the subacromial space, the patients were instructed to perform home physical therapy and follow-up in four weeks. Each patient was evaluated in terms of arc of motion, Visual Analog Scale and the UCLA Shoulder Rating Scale.

The outcome measures were taken at the preinjection state, immediately post injection, and at 4 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Shoulder pain characteristic of subacromial impingement syndrome with passive and/or active abduction in the 60-120 arc of motion (positive impingement sign)
2. Diagnosis of subacromial bursitis based on tenderness to palpation anterior/lateral to the acromion. Pain may be exacerbated with the shoulder held in internal rotation (positive Hawkins test)

Exclusion Criteria:

1. Age <18 years
2. Symptoms less than one month
3. Previous shoulder injections within the past 3 months
4. Evidence of os-acromiale or other confounding shoulder pathology on plain radiographs
5. Evidence of shoulder osteoarthritis
6. Full thickness rotator cuff tear evidenced by MRI, cuff weakness after lidocaine injection, or positive drop-arm sign
7. Systemic inflammatory condition
8. Pending litigation or work-related claims related to the shoulder
9. Previous shoulder surgery on the affected shoulder
10. Evidence of local infection
11. Evidence of adhesive capsulitis
12. Previous history of gastrointestinal ulcers or bleeding disorders
13. Evidence of shoulder instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
UCLA Shoulder Rating Scale | 4 Weeks
  This scoring system consists of subjective assessments of pain, function and satisfaction, as well as objective measurements of active forward elevation and strength in forward flexion.

SECONDARY OUTCOMES:
Visual Analog Scale | 4 Weeks
  This is a pain scale.
Range of Motion | 4 Weeks
  Shoulder Range of Motion was assessed with a hand held goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Kyong S Min, MD, Principal Investigator — Madigan Army Medical Center

REFERENCES:
- [Derived] Min KS, St Pierre P, Ryan PM, Marchant BG, Wilson CJ, Arrington ED. A double-blind randomized controlled trial comparing the effects of subacromial injection with corticosteroid versus NSAID in patients with shoulder impingement syndrome. J Shoulder Elbow Surg. 2013 May;22(5):595-601. doi: 10.1016/j.jse.2012.08.026. Epub 2012 Nov 22. PMID 23177167